CLINICAL TRIAL: NCT06201598
Title: Prospective, Single-Arm, Multicenter Study to Evaluate the Effectiveness and Safety of Endovascular Treatment in Patients With Cerebral Aneurysms Using P64 and P48 Flow-Diverter Stents
Acronym: pSPAIN_HPC
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario Central de Asturias (Other)
Responsible Party: Principal Investigator, Pedro Vega Valdes, PEDRO VEGA VALDES, Hospital Universitario Central de Asturias
Other Study IDs: 2023.014
Record Dates: First submitted 2023-12-15; First posted 2024-01-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Aneurysm; Thromboembolic Disease
Keywords: Cerebral aneurysm; Flow-diverting stents; Thrombogenicity; p64 MW HPC; p48 MW HPC
MeSH Terms: conditions — Intracranial Aneurysm; Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with p64MW HPC and p48MW HPC: Patients with intracranial aneurysms or dissections undergoing endovascular treatment with p64MW HPC and p48MW HPC flow-diverting devices.
  Interventions: Device: Group 1 - Intervention 1

INTERVENTIONS:
Device: Group 1 - Intervention 1 — Endovascular treatment of cerebral aneurysms through the implantation of p64MW HPC and p48MW HPC devices.

SUMMARY:
The use of flow-diverting stents for the endovascular treatment of cerebral aneurysms has proven to be effective and efficient in several clinical studies, leading to its widespread adoption. Devices with a higher number of filaments have a greater flow-diverting effect and less variation when there are changes in the caliber of the underlying vessel or in curved vessels. However, ischemic complications secondary to their implantation have been reported, prompting the development of various strategies to reduce their thrombogenicity. Phenox is the only company to date that has developed an anti-thrombogenic coating, known as HPC (Hydrophilic Polymer Coating), which, when applied to the p64 MW HPC and p48 MW HPC devices, has shown to reduce the likelihood of thromboembolic complications associated with their implantation.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effectiveness and safety of endovascular treatment for cerebral aneurysms using the flow-diverting stents p64MW (flow modulation device) HPC and p48MW HPC in the routine clinical practice of several Spanish hospitals. It is therefore an observational study, carried out with devices already commercialized. The success rate of the intervention, the rate of hemorrhagic and thromboembolic complications, as well as variables related to the clinical and radiological follow-up of patients over a 12-month period, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with incidental, symptomatic, and/or ruptured cerebral aneurysms.
* Signed informed consent by the patient or their representative.

Exclusion Criteria:

* Patients under 18 years of age.
* Absence of signed informed consent by the patient or their representative.
* Known, medically untreatable allergy to iodinated contrast.
* Pregnant women or those breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients with intracranial aneurysms or dissections suitable for endovascular treatment with a flow-diverting device, who attend the participating hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness objective | 1 year
  Evaluation of the effectiveness of treating cerebral aneurysms with p64MW HPC and p48MW HPC devices in several Spanish hospitals.
Safety Objective | 1 year
  Evaluation of the safety of treating cerebral aneurysms with p64MW HPC and p48MW HPC devices in several Spanish hospitals.

SECONDARY OUTCOMES:
Intervention success | During the procedure
  Rate of the ability to position the stent in the indicated location.
Thromboembolic complications | 1 year
  Rate of cerebral thromboembolic complications during the intervention and during patient follow-up.
Hemorrhagic complications | 1 year
  Rate of cerebral and systemic hemorrhagic complications during the intervention and during patient follow-up.
Mortality | 1 year
  Mortality rate during patient follow-up.
Clinical evolution of the patient using the National Institutes of Health Stroke Scale (NIHSS) and the Modified Rankin Scale (MRS). | 1 year
  NIHSS at 24 hours and at discharge (range 0-42, with higher scores indicating greater stroke severity).
  MRS at 24 hours, at discharge, at 4-6 months and 12 months post-treatment (range 0-6, from no symptoms to dead, for the evaluation of neurological functional disability).
Intimal hyperplasia | 1 year
  Rate of intimal hyperplasia within the stent leading to a luminal stenosis of over 50%, assessed through digital angiography at 4-6 months and 12 months post-treatment.
Thromboembolic complications with a single antiplatelet drug | 1 year
  Rate of thromboembolic complications during the intervention and patient follow-up in cases where a single antiplatelet drug is administered.
Intimal hyperplasia with a single antiplatelet drug | 1 year
  Rate of intimal hyperplasia within the stent leading to a luminal stenosis of over 50% in cases where a single antiplatelet drug is administered, assessed through digital angiography at 4-6 months and 12 months post-treatment.
Visible ischemic complications | 6 months
  Rate of visible ischemic complications in MRI during patient follow-up (4-6 months).
Aneurysm occlusion | 1 year
  Aneurysm occlusion rate assessed through digital angiography at 6 and 12 months post-intervention, according to the O'Kelly-Marotta (OKM) occlusion scale.

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Parc Tauli, Sabadell
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kallmes DF, Ding YH, Dai D, Kadirvel R, Lewis DA, Cloft HJ. A new endoluminal, flow-disrupting device for treatment of saccular aneurysms. Stroke. 2007 Aug;38(8):2346-52. doi: 10.1161/STROKEAHA.106.479576. Epub 2007 Jul 5. PMID 17615366
- [Background] Kadirvel R, Ding YH, Dai D, Rezek I, Lewis DA, Kallmes DF. Cellular mechanisms of aneurysm occlusion after treatment with a flow diverter. Radiology. 2014 Feb;270(2):394-9. doi: 10.1148/radiol.13130796. Epub 2013 Oct 28. PMID 24086073
- [Background] Cancelliere NM, Nicholson P, Radovanovic I, Mendes KM, Orru E, Krings T, Pereira VM. Comparison of intra-aneurysmal flow modification using optical flow imaging to evaluate the performance of Evolve and Pipeline flow diverting stents. J Neurointerv Surg. 2020 Aug;12(8):814-817. doi: 10.1136/neurintsurg-2019-015696. Epub 2020 Apr 21. PMID 32317371
- [Background] Shapiro M, Raz E, Becske T, Nelson PK. Variable porosity of the pipeline embolization device in straight and curved vessels: a guide for optimal deployment strategy. AJNR Am J Neuroradiol. 2014 Apr;35(4):727-33. doi: 10.3174/ajnr.A3742. Epub 2013 Sep 26. PMID 24072622
- [Background] Briganti F, Leone G, Marseglia M, Cicala D, Caranci F, Maiuri F. p64 Flow Modulation Device in the treatment of intracranial aneurysms: initial experience and technical aspects. J Neurointerv Surg. 2016 Feb;8(2):173-80. doi: 10.1136/neurintsurg-2015-011743. Epub 2015 Apr 20. PMID 25895510
- [Background] Fischer S, Aguilar-Perez M, Henkes E, Kurre W, Ganslandt O, Bazner H, Henkes H. Initial Experience with p64: A Novel Mechanically Detachable Flow Diverter for the Treatment of Intracranial Saccular Sidewall Aneurysms. AJNR Am J Neuroradiol. 2015 Nov;36(11):2082-9. doi: 10.3174/ajnr.A4420. Epub 2015 Aug 13. PMID 26272970
- [Background] Morais R, Mine B, Bruyere PJ, Naeije G, Lubicz B. Endovascular treatment of intracranial aneurysms with the p64 flow diverter stent: mid-term results in 35 patients with 41 intracranial aneurysms. Neuroradiology. 2017 Mar;59(3):263-269. doi: 10.1007/s00234-017-1786-2. Epub 2017 Feb 24. PMID 28236050
- [Background] Briganti F, Leone G, Ugga L, Marseglia M, Macera A, Manto A, Delehaye L, Resta M, Resta M, Burdi N, Nuzzi NP, Divenuto I, Caranci F, Muto M, Solari D, Cappabianca P, Maiuri F. Mid-term and long-term follow-up of intracranial aneurysms treated by the p64 Flow Modulation Device: a multicenter experience. J Neurointerv Surg. 2017 Jan;9(1):70-76. doi: 10.1136/neurintsurg-2016-012502. Epub 2016 Jul 20. PMID 27439887
- [Background] Aguilar Perez M, Henkes E, Hellstern V, Serna Candel C, Wendl C, Bazner H, Ganslandt O, Henkes H. Endovascular Treatment of Anterior Circulation Aneurysms With the p64 Flow Modulation Device: Mid- and Long-Term Results in 617 Aneurysms From a Single Center. Oper Neurosurg. 2021 Mar 15;20(4):355-363. doi: 10.1093/ons/opaa425. PMID 33469666
- [Background] De Beule T, Boulanger T, Heye S, van Rooij WJ, van Zwam WH, Stockx L. p64 flow diverter: Results in 108 patients from a single center. Interv Neuroradiol. 2021 Feb;27(1):51-59. doi: 10.1177/1591019920932048. Epub 2020 Jun 6. PMID 32506988
- [Background] Aguilar Perez M, Bhogal P, Henkes E, Ganslandt O, Bazner H, Henkes H. In-stent Stenosis after p64 Flow Diverter Treatment. Clin Neuroradiol. 2018 Dec;28(4):563-568. doi: 10.1007/s00062-017-0591-y. Epub 2017 May 9. PMID 28488025
- [Background] Sirakov S, Sirakov A, Bhogal P, Penkov M, Minkin K, Ninov K, Hristov H, Karakostov V, Raychev R. The p64 Flow Diverter-Mid-term and Long-term Results from a Single Center. Clin Neuroradiol. 2020 Sep;30(3):471-480. doi: 10.1007/s00062-019-00823-y. Epub 2019 Aug 9. PMID 31399749
- [Background] Bonafe A, Perez MA, Henkes H, Lylyk P, Bleise C, Gascou G, Sirakov S, Sirakov A, Stockx L, Turjman F, Petrov A, Roth C, Narata AP, Barreau X, Loehr C, Berlis A, Pierot L, Mis M, Goddard T, Clifton A, Klisch J, Walesa C, Dall'Olio M, Spelle L, Clarencon F, Yakovlev S, Keston P, Nuzzi NP, Dima S, Wendl C, Willems T, Schramm P. Diversion-p64: results from an international, prospective, multicenter, single-arm post-market study to assess the safety and effectiveness of the p64 flow modulation device. J Neurointerv Surg. 2022 Sep;14(9):898-903. doi: 10.1136/neurintsurg-2021-017809. Epub 2021 Nov 15. PMID 34782399
- [Background] Tonetti DA, Jankowitz BT, Gross BA. Antiplatelet Therapy in Flow Diversion. Neurosurgery. 2020 Jan 1;86(Suppl 1):S47-S52. doi: 10.1093/neuros/nyz391. PMID 31838537
- [Background] Lenz-Habijan T, Bhogal P, Peters M, Bufe A, Martinez Moreno R, Bannewitz C, Monstadt H, Henkes H. Hydrophilic Stent Coating Inhibits Platelet Adhesion on Stent Surfaces: Initial Results In Vitro. Cardiovasc Intervent Radiol. 2018 Nov;41(11):1779-1785. doi: 10.1007/s00270-018-2036-7. Epub 2018 Jul 23. PMID 30039502
- [Background] Hellstern V, Aguilar Perez M, Henkes E, Donauer E, Wendl C, Bazner H, Ganslandt O, Henkes H. Use of a p64 MW Flow Diverter with Hydrophilic Polymer Coating (HPC) and Prasugrel Single Antiplatelet Therapy for the Treatment of Unruptured Anterior Circulation Aneurysms: Safety Data and Short-term Occlusion Rates. Cardiovasc Intervent Radiol. 2022 Sep;45(9):1364-1374. doi: 10.1007/s00270-022-03153-8. Epub 2022 May 13. PMID 35562486